CLINICAL TRIAL: NCT04828629
Title: Complications and the Influence of COVID-19 on Myocardial Function and Exercise Capacity
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Polish Mother Memorial Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PMMHRI-BCO.75/2020
Record Dates: First submitted 2021-03-12; First posted 2021-04-02 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2023-11

CONDITIONS: Covid19; Heart Failure
MeSH Terms: conditions — COVID-19; Heart Failure | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Identification of prognostic factors in patients who have recovered from COVID-19: Selected prognosis factors will be analyzed in patients who have recovered from COVID-19
  Interventions: Diagnostic Test: Diagnostic tests

INTERVENTIONS:
Diagnostic Test: Diagnostic tests — Selected prognostic factors will be analyzed, among others: demographic data of the patient, physical examination, symptoms, co-morbidities, results of selected laboratory tests, lung imaging (X-ray or computed tomography) selected electrocardiographic and echocardiographic data, patient's cooperation with the doctor, treatment applied, parameters in the spiroergometric study, body mass analysis.

SUMMARY:
The subject of the study is the impact of COVID-19 on the indicators of myocardial efficiency and exercise capacity. As a result of the observed dependencies, it will be possible to start an appropriate diagnostic procedure early, select personalized treatment and develop a model of cardiological care for people with a history of SARS-CoV-2 infection and improve the quality and extend their life.

DETAILED DESCRIPTION:
About 100 adult patients hospitalized in the Department of Cardiology and Congenital Heart Diseases of Adults who had recovered from COVID-19 will be included in the study. Selected prognostic factors will be analyzed, among others: demographic data of the patient, physical examination, symptoms, co-morbidities, results of selected laboratory tests, lung imaging (X-ray or computed tomography) selected electrocardiographic and echocardiographic data, patient's cooperation with the doctor, treatment applied, parameters in the spiroergometric study, body mass analysis. One year after inclusion in the study, a control hospitalization will be performed. The same factors will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or older than 18 years
* infection with the SARS-CoV-2 in past medical history
* current hospitalization

Exclusion Criteria:

* severe hypertension;
* unstable angina;
* acute pulmonary embolism;
* decompensated heart failure;
* recent myocardial infarction;
* unstable heart rhythm disturbances;
* acute myocarditis or pericarditis;
* active endocarditis;
* advanced atrioventricular block;
* diagnosis of cardiomyopathy (hypertrophic, dilated, restrictive, peripartum, arrhythmogenic)
* lysosomal storage disorders
* severe hyper- and hypothyroidism
* pregnancy and lactation
* chronic kidney disease (IV, V stadium according to NKF) and dialysis treatment
* documented neoplastic process
* the patient's inability to cooperate and/or provide informed consent to participate in a research
* alcohol and drug abuse
* active autoimmune disease
* treatment using immunosuppressants, cytostatic drugs, glucocorticosteroids, or antiretroviral drugs
* a history of bone marrow transplant or other organ transplant, treatment with blood products within the last 6 months
* active systemic infection
* HBV, HCV or HIV carrier or positive for HbS antigen or antibodies to HCV
* surgery or serious injury within the last month
* patients who did not express their informed consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The 100 consecutive adult patients (18 years of age or older) hospitalized in the Department of Cardiology and Congenital Heart Diseases of Adults who had recovered from COVID-19 will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-12-23 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Prognosis in patients who have recovered from COVID-19 | 12 months after inclusion in the study
  A control hospitalization will be conducted with patients. The same prognostic factors will be analyzed: physical examination, symptoms, co-morbidities, treatment applied, results of selected laboratory tests, lung imaging (X-ray or computed tomography) selected electrocardiographic (ECG) and echocardiographic data, parameters in the spiroergometric study, body mass analysis.

SECONDARY OUTCOMES:
Review of selected laboratory tests in patients who have recovered from COVID-19 | 12 months after inclusion in the study
  Diagnostic blood samples will be collected from each patient: N-terminal pro b-type natriuretic peptide (NT-proBNP) and high sensitive cardiac Troponin T (hsTnT), the alanine aminotransferase (ALT) and aspartate transaminase (ASP), creatinine, glomerular filtration rate (GFR) estimate by Modification of Diet in Renal Disease (MDRD) parameters, inflammatory cytokine [C-reactive protein (CRP)], glucose level, lipoprotein profile: low density lipoprotein (LDL), high density lipoprotein (HDL), triglycerides (TG) and total cholesterol (TC). Also, the amount of hemoglobin will be performed.
The imaging of pulmonary changes in patients who have recovered from COVID-19 | 12 months after inclusion in the study
  Chest X-ray or lung computed tomography will be performed.
Review of selected Holter ECG monitoring data in patients who have recovered from COVID-19 | 12 months after inclusion in the study
  Analysis of average heart rate, ST segment abnormality (elevation or depression), the presence of: atrioventricular delay (AV block), bundle branch block, supraventricular and ventricular extrasystoles, atrial fibrillation (AF).
Review of selected echocardiographic data in patients who have recovered from COVID-19 | 12 months after inclusion in the study
  Measurement of left ventricular (LV) volume and ejection fraction (EF), left atrial (LA) volume, LA volume index (LAVi), maximal early (E) and late (A) transmitral velocities, ratio of early transmitral peak velocity to early diastolic peak annular velocity (E/E'), early diastolic (E'), late diastolic (A') mitral annular myocardial velocity of the left ventricle, LAVi/A', tricuspid annular plane systolic excursion (TAPSE).
Review of parameters in the spiroergometric study in patients who have recovered from COVID-19 | 12 months after inclusion in the study
  Forced vital capacity (FVC),forced expiratory volume in one second (FEV1), FEV1/FVC ratio, VO2max (represents the maximal achievable level of oxidative metabolism involving large muscle groups), ventilatory exchange (VE), oxygen uptake (VO2), CO2 expenditure (VCO2), respiratory exchange ratio (RER), anaerobic threshold (AT), oxygen uptake at anaerobic threshold (VO2 AT), the minute ventilation/carbon dioxide production slope (VE/VCO2 slope) will be performed.
Body mass analysis in patients who have recovered from COVID-19 | 12 months after inclusion in the study
  Body composition measurement will be conducted using bioelectrical impedance analysis (BIA). Fat mass (FM) and fat-free mass (FFM), total body water (TBW), extra-cellular (ECW) and intra-cellular (ICW) water, ECW/TBWx100% will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Agata Bielecka-Dabrowa, Study Chair — Heart Failure Unit; Department of Cardiology and Congenital Diseases of Adults, PMMHRI; Maciej Banach, Study Chair — Heart Failure Unit; Department of Cardiology and Congenital Diseases of Adults, PMMHRI
Locations (1):
- Heart Failure Unit; Department of Cardiology and Congenital Diseases of Adults, Polish Mother's Memorial Hospital Research Institute, Lodz, Polska, Poland

REFERENCES:
- [Derived] Gryglewska-Wawrzak K, Sakowicz A, Banach M, Bytyci I, Bielecka-Dabrowa A. Diagnostic Usefulness of Spiroergometry and Risk Factors of Long COVID in Patients with Normal Left Ventricular Ejection Fraction. J Clin Med. 2023 Jun 20;12(12):4160. doi: 10.3390/jcm12124160. PMID 37373853
- [Derived] Gryglewska-Wawrzak K, Sakowicz A, Banach M, Maciejewski M, Bielecka-Dabrowa A. Factors of Persistent Limited Exercise Tolerance in Patients after COVID-19 with Normal Left Ventricular Ejection Fraction. Biomedicines. 2022 Dec 15;10(12):3257. doi: 10.3390/biomedicines10123257. PMID 36552013